CLINICAL TRIAL: NCT05174468
Title: Analysis of Volatile Chemicals in Lung Cancer Screen-Eligible Subjects Using Infrared Spectroscopy
Status: Terminated | Type: Observational
Why Stopped: Change in sponsor's business strategy (disease focus changed to breast cancer)
Sponsor: Breathe BioMedical Inc (Industry)
Collaborators: West Virginia University (Other)
Responsible Party: Sponsor
Other Study IDs: WVU010521
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Lung Cancer
Keywords: Breath Analysis; Volatile Organic Compounds; Infrared Spectroscopy
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Volatile organic compounds (VOC) in breath are organic chemicals that are diffused or suspended at a room temperature. Breath samples will be collected into sorbent tubes that will be placed immediately (within ten minutes) after collection and stored in a freezer maintained at -1 to -10 degrees Fahrenheit and shipped on to Picomole headquarters for volatile chemical analysis using infrared spectroscopy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Screen-eligible Subjects: High-risk for lung cancer population who meet the USPSTF eligibility. One 10-L breath sample will be collected from each subject. During breath collection, subjects will be asked to exhale into a portable breath sampling device through a single use filter. Subjects will not be contacted to donate additional/serial breath specimens after the initial breath samples. Subjects will fill out a medical questionnaire and medical records will also be reviewed to extract low-dose CT scan (LDCT) screening results and any additional tumour-related information including histologic subtype, tumor stage, and sites of disease.

SUMMARY:
The aim of this study is to sample and analyze volatile organic compounds (VOCs) from a high-risk population of subjects eligible for lung cancer screening as defined by the US Preventive Services Task Force (USPSTF) guidelines. The breath sample analysis will help investigators describe and identify real-world breath profiles from individuals at high risk of developing lung cancer and to use this to test machine learning (ML) algorithms for lung cancer screening. This study will also evaluate the feasibility and usability of Picomole's breath sampling technology in a mobile platform.

with lung cancer when compared to normal breath profiles using infrared spectroscopy. This work will help validate early proof of concept results conducted with prototype technology and later stage NSCLC breath samples, and inform future breath testing analysis.

DETAILED DESCRIPTION:
Lung cancer is the most common malignancy in the world in terms of both incidence and mortality (1.1 million new cases per year and 0.95 million deaths in males and 0.51 million new cases per year and 0.43 million deaths in females). The highest rates of lung cancer are found in Europe and North America. In addition, lung cancer is the leading cause of cancer death in Canada. Lung cancer is believed to develop slowly via a progressive accumulation of genetic mutations, hence the disease allows time for diagnosis and curative surgical treatment. When detected in the early stages, the 5-year survival rate for NSCLC is 57% to 61%, compared with a survival rate of approximately 6% once distant metastases are present. Unfortunately, most patients do not experience any signs or symptoms of lung cancer until the disease has progressed to an advanced stage. Therefore, technologies that facilitate detection of lung cancer in the earliest asymptomatic stages have significant potential to reduce lung cancer-specific mortality.

Malignant transformation is facilitated by deregulation of fundamental cellular processes, including alterations in metabolism. Thus, metabolomic profiling may be a promising strategy for identifying lung cancer before it is detectable via conventional methods such as CT scans. Breathomics is a field of study dedicated to deconstructing the metabolomic profile or biological components of volatile organic compounds (VOC) in breath. To date, various analytical techniques including gas chromatography combined with mass spectrometry, ion mobility spectrometry, proton transfer reaction spectrometry, and selected ion flow tube mass spectrometry have been used to study breath VOCs. In a recent study, ion mobility spectrometry discriminated between lung cancer and chronic obstructive lung disease with 79% accuracy, 76.8% sensitivity, and 85.7% specificity. Furthermore, breath analysis can be used to not only identify lung cancer but also distinguish between lung cancers with particular somatic mutations. For example, electronic nose technology demonstrated 79% and 85% sensitivity and specificity, respectively, for identifying EGFR-mutant lung cancer. These studies suggest that breath analysis is a highly sensitive and specific approach to detecting lung cancer.

This study will evaluate the performance characteristics of infrared spectroscopy for breath analysis. The spectrometer used to analyze breath gases is optimized to measure chemical concentrations down to the parts per trillion range. In a pilot study of 165 (67 newly diagnosed Non-Small Cell Lung Cancer (NSCLC) subjects which used infrared spectroscopy to analyze breath specimens from subjects with lung cancer and subjects without cancer, sensitivity and specificity for detecting lung cancer was 88.7% and 80%, respectively, with an accuracy of 86%. These preliminary results compare very favorably to mass spectrometry (the analytical platform that has been used in most breath analysis studies).

This study will analyze breath VOCs from 300 subjects who meet the USPSTF eligibility guidelines for lung cancer screening. The study aims to better understand the VOC breath profiles in a larger group of subjects at high risk for developing lung cancer. By restricting the population to screen-eligible subjects, this study will approximate the potential future "real world" use of this screening strategy and better approximate its utility in the field, sampling high risk populations in rural settings. It is envisioned that this study will generate preliminary data that will inform the performance of machine learning algorithms developed to detect the presence of lung cancer in unselected populations.

ELIGIBILITY:
Inclusion Criteria:

* Being screened for lung cancer on LUCAS;
* At high-risk for lung cancer based on USPSTF guidelines:
* Asymptomatic adults aged 50-80 years
* Tobacco smoking history of at least 20 pack-years (one pack-year = smoking one pack per day for one year; 1 pack = 20 cigarettes)
* Current smoker or has quit smoking within the past 15 years.
* No history of lung cancer or any other active cancer within 3 years (Note: DCIS, CIN, non-invasive bladder cancer, non-melanomatous skin cancers are an exception);
* Ability to provide a breath sample;
* Ability to give informed consent.

Exclusion Criteria:

* Persons who cannot give informed consent or assent (i.e. mentally incompetent persons, or those physically incapacitated) or do not have a legally acceptable representative are not to be recruited into this study;
* Persons who require the use of supplemental oxygen;
* The breath sampling technology is sensitive to the chemicals produced by tobacco, cannabis, and e-cigarettes as well as alcohol (consumed by the subject or used by the operator around the equipment). So we ask that subjects refrain from Smoking (tobacco, cannabis, or e-cigarettes ) at least 4 hours before and consuming alcohol (including mouthwash) 8 hours before breath sampling

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects who meet the USPSTF eligibility guidelines for lung cancer screening
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-07-12 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
VOC spectral profile differences | within 30 days after collection
  VOC spectral profiles will be compared between cohorts to identify statistical differences

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Chapman, MD, Principal Investigator — West Virginia University , Department of Medicine
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Boots AW, van Berkel JJ, Dallinga JW, Smolinska A, Wouters EF, van Schooten FJ. The versatile use of exhaled volatile organic compounds in human health and disease. J Breath Res. 2012 Jun;6(2):027108. doi: 10.1088/1752-7155/6/2/027108. Epub 2012 May 23. PMID 22621865
- [Background] Shlomi D, Abud M, Liran O, Bar J, Gai-Mor N, Ilouze M, Onn A, Ben-Nun A, Haick H, Peled N. Detection of Lung Cancer and EGFR Mutation by Electronic Nose System. J Thorac Oncol. 2017 Oct;12(10):1544-1551. doi: 10.1016/j.jtho.2017.06.073. Epub 2017 Jul 12. PMID 28709937
- [Background] Schmidt FM, Metsala M, Vaittinen O, Halonen L. Background levels and diurnal variations of hydrogen cyanide in breath and emitted from skin. J Breath Res. 2011 Dec;5(4):046004. doi: 10.1088/1752-7155/5/4/046004. Epub 2011 Aug 2. PMID 21808098
- [Background] Chen W, Metsala M, Vaittinen O, Halonen L. Hydrogen cyanide in the headspace of oral fluid and in mouth-exhaled breath. J Breath Res. 2014 Jun;8(2):027108. doi: 10.1088/1752-7155/8/2/027108. Epub 2014 May 21. PMID 24844251
- See also: American Cancer Society. Cancer Facts & Figures 2019. Atlanta: American Cancer Society — https://www.cancer.org/research/cancer-facts-statistics/all-cancer-facts-figures/cancer-facts-figures-2019.html
- See also: Canadian Cancer Statistics 2019 — https://cdn.cancer.ca/-/media/files/research/cancer-statistics/2019-statistics/canadian-cancer-statistics-2019-en.pdf
- See also: The American Cancer Society (2016). Non-Small Cell Lung Cancer Survival Rates. — https://www.cancer.org/cancer/lung-cancer/detection-diagnosis-staging/survival-rates.html
- See also: [Abstract] Janssens E, Lamote K, van Meerbeeck JP (2018). Breath analysis by ion mobility spectrometry allows to discriminate COPD from lung cancer patients. European Respiratory Journal. 52: Suppl. 62, — http://www.owlstonemedical.com/media/uploads/files/Janssens-Breath_analysis_by_ion_mobility_spectrometry.pdf